CLINICAL TRIAL: NCT06884826
Title: Evaluation of Desarda Technique in Management of Complicated Inguinal Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mohamed Salah, Lecturer of General Surgery, Faculty of Medicine, Minia University, Minia, Egypt., Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1242/08/2024
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Desarda; Complicated; Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Desarda technique group (Experimental): Patients will undergo Desarda technique.
  Interventions: Procedure: Desarda technique

INTERVENTIONS:
Procedure: Desarda technique — Patients will undergo Desarda technique.

SUMMARY:
This study aims to evaluate the desarda technique in management of complicated inguinal hernia.

DETAILED DESCRIPTION:
Desarda technique is one of the best surgical methods suitable for emergency hernia surgery repair, but there is still limited consensus. The purpose of this study is to assess the Long-term outcome of the pure tissue Desarda technique for the treatment of emergency inguinal hernias repair (Incarcerated, Irreducible, and Obstructed Patients) regarding Postoperative Complications, Groin Pain, and recurrence rate.

Surgical techniques for emergency inguinal hernia surgery remain an important less documented area. Emergency inguinal hernia can have different presentations. Incarceration is characterized by the irreducibility of contents and strangulation by the compromise of the blood supply of the contents (e.g., bowel, omentum).

ELIGIBILITY:
Inclusion Criteria:

* Age above 14 years old.
* Irreducible, incarcerated & obstructed inguinal or inguinoscrotal hernia; unilateral or bilateral

Exclusion Criteria:

* Recurrent Hernias.
* Intra-operative finding of separated thin and/or weak external oblique aponeurosis.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative complications | 24 hours postoperatively
  Incidence of postoperative complications such as groin pain, hemorrhage, infection, seroma, orchitis, and testicular atrophy will be recorded.

SECONDARY OUTCOMES:
Stop of postoperative analgesic | 6 days postoperatively
  Stop of postoperative analgesic (Within 3 days, 3-6 day, More than 6 days) will be recorded.
Incidence of recurrence | 1 year postoperatively
  Incidence of recurrence will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.